CLINICAL TRIAL: NCT05946603
Title: Phase 2 Multi-Center Randomized Controlled Feasibility Study of IS-002 in Subjects Undergoing Robotic-Assisted Radical Prostatectomy Using the da Vinci® Surgical System With Firefly® Fluorescence Imaging
Brief Title: IS-002 Phase 2 Prostate Cancer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ISI-142325-2
Record Dates: First submitted 2023-06-28; First posted 2023-07-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RARP + IS-002 (Sham Comparator): Subjects will receive IS-002, but during surgery NO fluorescence imaging will be performed.
  Interventions: Drug: Administration of IS-002; Procedure: robotic-assisted laparoscopic prostatectomy with pelvic lymph node dissection
- RARP + IS-002 + intraoperative near-infrared imaging (Experimental): Subjects will receive IS-002, and during surgery fluorescence imaging will be performed.
  Interventions: Drug: Administration of IS-002; Device: Firefly fluorescent imaging; Procedure: robotic-assisted laparoscopic prostatectomy with pelvic lymph node dissection

INTERVENTIONS:
Drug: Administration of IS-002 — Intravenous administration of IS-002 approximately 24 hours prior to surgery
Device: Firefly fluorescent imaging — Near-infrared fluorescence imaging using Firefly technology will allow fluorescence imaging of IS-002
  Arms: RARP + IS-002 + intraoperative near-infrared imaging
Procedure: robotic-assisted laparoscopic prostatectomy with pelvic lymph node dissection — Subject will undergo robotic-assisted laparoscopic prostatectomy with pelvic lymph node dissection
  Other Names: RARP

SUMMARY:
Phase 2 randomized controlled multi-center study of IS-002, in conjunction with near-infrared (NIR) fluorescence imaging, for identification of prostate cancer during robotic-assisted radical prostatectomy (RARP) with (extended) pelvic lymph node dissection ((e)PLND) using the da Vinci® X/Xi Surgical System with Firefly® Fluorescence Imaging.

ELIGIBILITY:
Inclusion criteria

1. Subjects aged 18 to 75.
2. Subject has a confirmed adenocarcinoma of the prostate as defined by (histo-) pathology.
3. Subject has CAPRA ≥6; or ≥T3 disease on imaging (TRUS and/or MRI); or a Gleason sum score ≥8; or regional lymphadenopathy suspicious for nodal metastases on imaging.
4. Subject is scheduled to undergo robotic-assisted radical prostatectomy (RARP) with (extended) pelvic lymph node dissection ((e)PLND) using a da Vinci® X/Xi Surgical System equipped with Firefly® Fluorescence Imaging.
5. Subject is willing and able to provide written informed consent.
6. Subject can comply with the study procedures and study visits and understands an informed consent document.

Exclusion criteria

1. Subject has known bone metastasis.
2. Subject has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
3. Subject has a known history of acute or chronic liver or kidney disease.

   • Renal function at screening: i. Creatinine clearance: <50 mL/min as determined using the Cockcroft-Gault formula ii. Albumin: <LLN

   • Hepatic function at screening: i. AST and/or ALT: >2.5x ULN ii. Total Bilirubin (serum): >1.5x ULN
4. Subject has received neo-adjuvant therapy, radiation therapy, focal ablation therapy, hormonal therapy, or androgen deprivation therapy within the last 4 months.
5. Subject is currently receiving an investigational therapeutic agent; or has participated in a study of an investigational therapeutic agent within the past 6 months prior to the day of IS-002 infusion; or is involved in a significant risk investigational device study within the past 6 months prior to the day of IS-002 infusion.
6. Subject has any other condition or personal circumstance that, in the judgment of the site Investigator, might interfere with the collection of complete quality data or represents an unacceptable safety profile.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with ≥1 positive surgical margins (PSMs) on final histopathologic assessment in the Intervention arm and the Control arm. | Within 3 months post-surgery
  The proportion of subjects with ≥1 PSMs on final histopathologic assessment in the Intervention arm and the Control arm.
The mean number of positive surgical margins (PSMs) on final histopathologic assessment in the Intervention arm and the Control arm. | Within 3 months post-surgery
  The mean number of PSMs on final histopathologic assessment in the Intervention arm and the Control arm.

SECONDARY OUTCOMES:
Diagnostic performance of IS-002 fluorescence | Up to 1 year post-surgery
  The key secondary outcome is the determination of false-positive, true-positive, false-negative and true-negatives rates.
Safety: Adverse event assessment | Up to 1 year post-surgery
  Incidence of treatment-emergent adverse events from time of IS-002 administration through study exit using CTCAE v5.0
Pharmacokinetics: Area under the concentration-time curve (AUC) | Up to 24 hours post-IS-002 administration
  Area under the concentration-time curve (AUC) from time zero to the time of the last measurable concentration as calculated by linear up/log down trapezoidal method (AUC0-last)
Time to biochemical recurrence (BCR) | Up to 1 year post-surgery
  Time to BCR in the Intervention arm and the Control arm. BCR is defined a PSA level >0.1 ng/mL as determined by an ultrasensitive PSA assay.
Time to secondary treatment initiation | Up to 1 year post-surgery
  Time to secondary treatment(s) for prostate cancer in the Intervention arm and the Control arm.
Number of intraoperative fluorescent lymph nodes that are tumor positive that would not have been resected if the surgeon would have had access to white light imaging only | Up to 3 months post surgery
  In the Intervention arm, the number of intraoperative fluorescent lymph nodes, per subject and per lymph node basin, that are tumor positive that would not have been resected if the surgeon would have had access to white light imaging only.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCSF, San Francisco, California
  - Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - MSKCC, New York, New York

IPD SHARING:
Plan to Share IPD: No